CLINICAL TRIAL: NCT06005441
Title: A Phase 2b, Randomized, Placebo-Controlled Factorial Study to Evaluate the Efficacy, Safety and Tolerability of CBL-514 Injection Compared With CBL-A1 and CBL-A2 for Reducing Abdominal Subcutaneous Fat
Brief Title: A Phase 2b Study to Evaluate the Efficacy and Safety of CBL-514 Injection for Reducing Subcutaneous Fat.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBL-0205
Record Dates: First submitted 2023-08-10; First posted 2023-08-22 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Subcutaneous Fat
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CBL-514 Injection (Experimental): Participant will receive CBL-514 administered in 2.4 mL injections, up to 120 mL per treatment session at intervals of approximately 3 weeks for up to 4 treatments.
  Interventions: Drug: CBL-514 injection
- CBL-A1 Injection (Experimental): Participant will receive CBL-A1 administered in 2.4 mL injections, up to 120 mL per treatment session at intervals of approximately 3 weeks for up to 4 treatments.
  Interventions: Drug: CBL-A1 Injection
- CBL-A2 Injection (Experimental): Participant will receive CBL-A2 administered in 2.4 mL injections, up to 120 mL per treatment session at intervals of approximately 3 weeks for up to 4 treatments.
  Interventions: Drug: CBL-A2 Injection
- 0.9% Sodium Chloride (Placebo Comparator): Participant will receive 0.9% Sodium Chloride administered in 2.4 mL injections, up to 120 mL per treatment session at intervals of approximately 3 weeks for up to 4 treatments.
  Interventions: Drug: 0.9% Sodium Chloride

INTERVENTIONS:
Drug: CBL-514 injection — Provided as a ready for use injectable CBL-514 solution
  Arms: CBL-514 Injection
Drug: CBL-A1 Injection — Provided as a ready for use injectable CBL-A1 solution
  Arms: CBL-A1 Injection
Drug: CBL-A2 Injection — Provided as a ready for use injectable CBL-A2 solution
  Arms: CBL-A2 Injection
Drug: 0.9% Sodium Chloride — Sodium Chloride (0.9% NaCl) placebo for injection
  Arms: 0.9% Sodium Chloride

SUMMARY:
This is a randomized, placebo-controlled, Phase 2b study to evaluate the efficacy, safety, and tolerability of CBL-514 injection compared with CBL-A1 and CBL-A2 for reducing subcutaneous fat.

DETAILED DESCRIPTION:
A total of approximately 160 adult participants with moderate or severe abdominal fat at Screening will be enrolled. Each participant will receive up to 4 treatments of allocated study drug administered subcutaneously to the abdomen, once every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 years to 64 years old (at Screening), inclusive.
2. Body mass index (BMI) >18.5 and < 30 kg/m2 and body weight ≥ 50 kg at Screening and Day 1.
3. Participant has abdominal fat graded by the Investigator as Grade 3(moderate) or Grade 4(severe) using the Clinician-Reported Abdominal Fat Rating Scale at Screening.
4. Participant has stable body weight (identified as ≤ 3 kg weight change per participant report) for at least 3 months before Screening and during the study.
5. Participant who has maintained a stable lifestyle (e.g., exercise, eating patterns, and smoking habit) per participant report for at least 3 months before Screening and during the study.
6. Voluntarily signs the Informed Consent Form and, in the opinion of the Investigator or delegate, is physically and mentally capable of participating in the study and willing to adhere to study procedures.

Exclusion Criteria:

1. Female participant of childbearing potential who is not willing to commit to an acceptable contraceptive regimen from the time of Screening and throughout study participation until 90 days after the last IP dose, or who is currently pregnant or lactating. Male participant who is not willing to commit to using a condom and refraining from sperm donation from the time of the first dose of IP, throughout study participation until 90 days after the last IP dose.
2. Participant diagnosed with coagulation disorders or who is receiving anticoagulant/antiplatelet therapy or medications or dietary supplements that impede coagulation or platelet aggregation.
3. Participant has hemoglobin A1c (HbA1c) ≥9%, delayed wound healing, or poorly controlled diabetes in the opinion of Investigator, make the individual an inappropriate candidate for the study.
4. Participant with active or prior history of malignancies within 5 years before Screening or currently being evaluated for a possible malignancy at Investigator's discretion.
5. Participant with a history of human immunodeficiency virus (HIV)-1 infection or active HIV infection at Screening with positive HIV antigen/antibody combo test.
6. Participant with a history of trypanophobia, the extreme fear of medical procedures involving injections or needles, or who experiences vasovagal syncope or faints at the sight of blood or a needle.
7. Participant with folding fat or skin on abdomen in standing position.
8. Participant with severe or very severe abdominal visceral fat.
9. Participant with ventral abdominal or umbilical hernia or previous repair of same.
10. Participant has abnormal skin or local skin conditions at the treatment area, which, in the opinion of Investigator, would increase risk to the participant or inhibit safety and efficacy evaluation.
11. Participant who has undergone the following procedures:

    1. Previous surgery that caused scar tissues on the anticipated treatment area before Screening or during the study.
    2. Liposuction or abdominoplasty to the region to be treated before Screening or during the study.
    3. Aesthetic procedure for body contouring or fat reduction to the region to be treated within 12 months before Screening or during the study.
    4. Using medication that is delivered via subcutaneous injection at the treatment area within 4 weeks before Screening or during the study.
12. Participant with contraindications to MRI imaging
13. Participant is on prescription or OTC weight reduction medication, weight reduction program, or any GLP-1 agonist (e.g., semaglutide, terzepatide, liraglutide, etc.) (oral or injectable) within 6 months before Screening or during the study.
14. Participant is undergoing chronic steroid or immunosuppressive therapy.
15. Requiring continual use of any medication that is known to strongly inhibit or induce CYP1A2 enzymes, sensitive CYP1A2 substrates or drugs with narrow therapeutic index during the study that, in the opinion of the Investigator, may affect the evaluation of the study product or place the participant at undue risk.
16. Unable to receive local anesthesia.
17. Participant with known allergies or sensitivities to the IP or its components.
18. Participant with liver cirrhosis, with inadequate liver function at Screening.
19. Participant with any renal impairment.
20. Use of any investigational drug or device within 3 months prior to Screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with at least 20% subcutaneous fat change compared to Baseline, of CBL-514 compared with placebo | From Baseline to 4 weeks after the final treatment
  Measured by MRI

SECONDARY OUTCOMES:
Percentage of participants with at least 20% subcutaneous fat change compared to Baseline, of CBL-514 compared with CBL-A1 and CBL-A2 | From Baseline to 4 weeks after the final treatment
  Measured by MRI
Participants with at least 1-grade improvement reported by the Investigator using the Clinician-Reported Abdominal Fat Rating Scale (CR-AFRS) | From Baseline to 4 weeks after the final treatment
  The scale is a 5-point ordinal scale to assess the abdominal fat level
Participants with at least 2-grade improvement reported by the Investigator using the Clinician-Reported Abdominal Fat Rating Scale (CR-AFRS) | From Baseline to 4 weeks after the final treatment
  The scale is a 5-point ordinal scale to assess the abdominal fat level
Participants with at least 1-grade improvement reported by the participant using the Patient-Reported Abdominal Fat Rating Scale (PR-AFRS) | From Baseline to 4 weeks after the final treatment
  The scale is a 5-point ordinal scale to assess the abdominal fat level
Participants with at least 2-grade improvement reported by the participant using the Patient-Reported Abdominal Fat Rating Scale (PR-AFRS) | From Baseline to 4 weeks after the final treatment
  The scale is a 5-point ordinal scale to assess the abdominal fat level

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sheu, Study Director — Caliway Biopharmaceuticals Co., Ltd.
Locations (1):
- Investigational Site 1, Omaha, Nebraska, United States